CLINICAL TRIAL: NCT07357090
Title: Mechanisms Underlying Carbon Dioxide Induced Protein Efflux in Health and Traumatic Brain Injury
Brief Title: Carbon Dioxide Administration and Brain Waste Clearance
Acronym: COPETBI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew Mayer (Other)
Responsible Party: Sponsor-Investigator, Andrew Mayer, Professor of Translational Research, The Mind Research Network
Organization: The Mind Research Network (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 25-415
Record Dates: First submitted 2026-01-09; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury; Aging Disorder; Magnetic Resonance Imaging (MRI)
Keywords: Traumatic Brain Injury; Magnetic Resonance Imaging
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individuals with TBI (Experimental): A counter-balanced, cross-over design (AB/BA), in which individuals with TBI (aged 18-82 years) may be dosed to achieve 5 or 10 mmHG changes in ETCO2 across multiple visits.
  Interventions: Other: Hypercapnia task performed during fMRI
- Healthy Subjects (Experimental): A counter-balanced, cross-over design (AB/BA), in which individuals without a history of TBI (healthy subjects, aged 18-82 years) may be dosed to achieve 5 or 10 mmHG changes in ETCO2 across multiple visits.
  Interventions: Other: Hypercapnia task performed during fMRI

INTERVENTIONS:
Other: Hypercapnia task performed during fMRI — This study looks at different levels of carbon dioxide (CO2) exposure (changes of approximately 5 or 10 mmHg) on the brain and proteins in blood, in response to a hypercapnia task while participants undergo MRI. This sequence will dynamically mix gases to target an increase of 5 or 10 mmHg in ETCO2 (increase of ~5-7% CO2 and equal decrease in nitrogen) while keeping O2 constant.

SUMMARY:
The current study tests whether different exposures to carbon dioxide (CO2) can safely result in the increased movement of proteins from the brain into the blood. The investigators believe that this would be a proxy for the brain clearing waste products more effectively. The current study will use a counter-balanced design, in which individuals with and without a history of traumatic brain injury (TBI) will receive different levels of CO2 (targeted changes of approximately 5 or 10 mmHG in end-tidal CO2) approximately one week apart. The counter-balanced design means that each participant receives a single dose of CO2 at each visit, and different doses of CO2 at each visit. The order in which participants receive the dose is randomized, and the participant will not be informed of the dose.

DETAILED DESCRIPTION:
Impaired clearance of metabolic waste and cellular debris is a hallmark of TBI and other neurodegenerative conditions. Clearance primarily occurs through glymphatic/lymphatic pathways, which is partially dependent on the influx of cerebrospinal fluid (CSF). CSF flow is greatest during sleep, when low-frequency oscillations in cerebral blood volume are most prominent. The investigators propose that changing levels of cerebral blood volume via the administration of CO2 will drive CSF flow and ultimately promote brain waste clearance. The proposed study is significant because it examines whether prescribed CO2 can enhance protein efflux (i.e., a surrogate for waste clearance), and the biological mechanisms that may mediate this mechanism in both health and disease. The first study aim is therefore to determine whether the administration of CO2, a potent vasodilator, can be prescribed to mimic global changes in cerebral blood volume in a dose-dependent fashion. Basal protein levels and efflux (i.e., change from baseline) are quantified using high-sensitivity proteomic platforms. The second aim is to examine how individual differences in cerebrovascular function and other disease factors such as atrophy affect CO2-induced protein efflux.

Using a counter-balanced (AB/BA) design, individuals (aged 18-82 years) with chronic TBI and individuals without a history of TBI (healthy subjects) will be dosed to achieve either 5 or 10 mmHG changes in end-tidal CO2. Importantly, the proposed cerebrovascular mechanisms and surrogate markers of waste clearance are readily quantified in humans using advanced MR-imaging and commercially available proteomic platforms, exponentially increasing their clinical translation.

ELIGIBILITY:
Inclusion criteria for TBI cohort: 1) Able to give valid informed consent, 2) 18-82 years old, 3) history of TBI of any severity level (mild, moderate or severe) that was sustained in adulthood (age 18 and older), which will be confirmed using a semi-structured identification method (includes asking about loss of consciousness, posttraumatic amnesia, and feeling dazed/confused).

Inclusion criteria for Healthy Subjects cohort: 1) Able to give valid informed consent and 2) 18-82 years old years old.

Exclusion criteria for TBI cohort: 1) contraindications to MRI scanning including pregnancy or claustrophobia, 2) unable to give valid informed consent, incarcerated, 3) diagnosed with Alzheimer's, ADRD or mild cognitive impairment, 4) pre-existing history of autism spectrum disorders, intellectual disability, serious neurological (e.g., epilepsy, tumors, other conditions requiring neurosurgery) or psychiatric disorders (requiring hospitalization) prior to TBI onset, 5) current or previous diagnosis of a psychosis spectrum disorder or bipolar disorder, 6) respiratory diseases or pulmonary conditions that may increase the risk of study procedures (e.g., severe asthma, chronic obstructive pulmonary disease or other significant respiratory disorders), 7) a history of cardiac arrythmias 8) history of a current substance use disorder, 9) non-English fluency (based on screener), 10) Weigh under 110 pounds for blood draw.

Exclusion criteria for Healthy Subjects cohort: 1) contraindications to MRI scanning including pregnancy or claustrophobia, 2) unable to give valid informed consent, incarcerated, 3) diagnosed with Alzheimer's, ADRD or mild cognitive impairment, 4) history of developmental, neurological, or psychiatric disorders requiring hospitalization, 5) regular use of any substance in the past six months (i.e., no current use confirmed with urine screening), 6) previous head injury with greater than 30 minutes loss of consciousness, 7) respiratory diseases or pulmonary conditions that may increase the risk of study procedures (e.g., severe asthma, chronic obstructive pulmonary disease or other significant respiratory disorders), 8) a history of cardiac arrythmias, 9) non-English fluency (based on screener), 10) Weigh under 110 pounds for blood draw.

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2032-02 (Estimated)

PRIMARY OUTCOMES:
Cerebrovascular Reactivity (CVR), vascular-elicited bulk cerebral spinal fluid (VE-bCSF) | 2.5 hours post-intervention. Data will be reported at the conclusion of the study for all participants.
  Cerebrovascular reactivity (CVR) will be quantified using time-shifted end-tidal carbon dioxide (ETCO₂) regressors to model blood oxygen level-dependent (BOLD) changes using functional magnetic resonance imaging, capturing the temporally lagged positive relationship between ETCO₂ and the BOLD signal. Vascular enhanced changes in bulk CSF flow will be assessed by regressing band-pass filtered global grey matter signals and their derivatives on CSF bulk flow to capture the temporally lagged, negative relationship. Both of these measurements are in arbitrary units, and will be quantified by calculating percent signal change and statistical fit between regressors.
Protein Efflux (Surrogate Measure of Brain Waste Clearance) | Blood will be drawn at baseline, immediately prior to hypercapnia, 45 minutes post-hypercapnia, 90 minutes post-hypercapnia and 150 minutes post-hypercapnia. Data will be reported at the conclusion of the study for all participants.
  Protein efflux from the brain to the blood will be measured using Quanterix platform, with primary proteins including neurofilament light chain, brain-derived tau and glial fibrillary acidic protein (units=picogram/milligram).
  For neurofilament light chain (NfL), the limit of detection (LOD) is 0.104 pg/mL, the range is 0.025-0.276 pg/mL, and the lower limit of quantification (LLOQ) is 0.241 pg/mL. For glial fibrillary acidic protein (GFAP), the LOD is 0.221 pg/mL, the range is 0.042-0.481 pg/mL, and the LLOQ is 0.467 pg/mL. For brain-derived tau (BD Tau), the LOD is 0.024 pg/mL, the range is 0.007-0.059 pg/mL, and the LLOQ is 0.053 pg/mL. All values are obtained from the Quanterix website datasheets.

SECONDARY OUTCOMES:
Cognitive functioning | Pre (15-20 minutes) and post (15-20 minutes) intervention. Data will be reported at the conclusion of the study for all participants.
  A Working Memory Multimodal Attention Task will be used to examine cognitive functioning. Auditory and visual cues are simultaneously presented on a black or a gray background, and a cue prompts participants to attend to either modality. Cues are followed by simultaneously presented congruent or incongruent numeric targets ("one", "two" or "three"). Participants press a button corresponding to the target in the attended modality while ignoring information in the unattended modality (black background). Reactive control is quantified via subtraction of congruent from incongruent trials (i.e., large difference=poor reactive control). Participants are required to hold the attended stimuli in working memory for 1.5 seconds while ignoring the other modality, and to only respond when the next trial appears during proactive control (1-back), quantified by subtracting congruent 0-back from congruent 1-back trial. Outcomes are accuracy (scale of 0-100%) and reaction time (unit=millisecond).
Symptoms | After the first blood draw (i.e., blood collected at baseline), 10 and 20 minutes post-hypercapnia, as well as after blood collected 90-minutes post-hypercapnia. Data will be reported at the conclusion of the study for all participants.
  Participants will be asked to rate 4 different symptoms (current headache, current dizziness, current nausea, and current fogginess) on a Likert scale (range 0-10 for each symptom) at multiple times during the study. Symptom ratings will be summed to create a single summary score that can range between 0 and 40.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Mayer, Phd, Principal Investigator — Mind Research Network
Locations (1):
- The Mind Research Network, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No